CLINICAL TRIAL: NCT00542529
Title: Phase I/II, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation, Single-Center Study of the Progenitor Cell Mobilizing Effects of Imprime PGG™ Injection Administered at Varied Dosing Regimens With G-CSF Versus G-CSF Alone in Healthy Subjects
Brief Title: Phase I/II, Randomized, Double-Blind, Study of the Progenitor Cell Mobilizing Effects of Imprime PGG™ Injection Administered at Varied Dosing Regimens With G-CSF Versus G-CSF Alone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BT-CL-PGG-SCM0611
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2007-10

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Placebo Comparator): Placebo or 2.0 mg/kg of Imprime PGG dosed in 7 different treatment regimens in combination with G-CSF for up to 4 consecutive days.
  Interventions: Biological: Imprime PGG TM for Injection
- Cohort 2 (Placebo Comparator): Placebo or 4.0 mg/kg of Imprime PGG dosed in 7 different treatment regimens in combination with G-CSF for up to 4 consecutive days.
  Interventions: Biological: Imprime PGG TM for Injection

INTERVENTIONS:
Biological: Imprime PGG TM for Injection — Doses of 2.0 and 4.0 mg/kg intravenous Imprime PGG administered over 1-2 hr for up to 4 consecutive days

SUMMARY:
This study is a randomized, placebo-controlled, dose-escalation, single-center study evaluating two different doses of Imprime PGG, each in 7 different dosing regimes. A total of 66 subjects will be enrolled into 2 cohorts and, within each cohort, randomized to 1 of 7 treatment groups receiving Imprime PGG or placebo in varied dosing regimens with granulocyte-colony stimulating factor (G-CSF).

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 45, inclusive
2. Have a body weight of 45 kg to 125 kg, inclusive, and a body mass index less than or equal to 30 kg/m2
3. Be healthy based on medical history, physical examination, electrocardiogram (ECG), and clinical laboratory test results
4. If female, be non-pregnant and non-nursing. For either gender, the subject must be either sexually inactive (14 days prior to the first dose of study drug and throughout the study) or practicing at least two methods of birth control from the following list of acceptable forms of contraception:

   1. Surgically sterile subject or partner (bilateral tubal ligation, hysterectomy, bilateral oophorectomy or vasectomy performed at least 6 months prior to first dose of study drug)
   2. Intrauterine device (IUD) in place for at least 3 months
   3. Barrier methods (condom, diaphragm) with spermicide from the time of the subject/partner's last menstrual period and throughout the study
   4. Hormonal contraceptives for at least 3 months prior to the first dose of study drug
5. Has read, understood and signed the IRB-approved informed consent form (ICF)

Exclusion Criteria:

1. Has a known hypersensitivity to baker's yeast, G-CSF, or E.coli-derived proteins, or has an active yeast infection
2. Has any clinical condition that, in the opinion of the investigator, warrants exclusion from the study from a scientific, procedural, or safety perspective
3. Has a history of tobacco use within 90 days of the last day of screening (Day -1) or be a known or suspected abuser of alcohol or other drugs/substances of abuse
4. Has a positive hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) test conducted as part of screening
5. Except as otherwise indicated, has taken any prescription medication within 30 days of the last day of screening (Day -1) or over-the-counter medication, herbal preparation, or vitamins within 7 days of the last day of screening (Day -1)
6. Has participated in an investigational drug study within 30 days or five half-lives (whichever is longer) of the last day of screening (Day -1), has received G-CSF within 30 days of the last day of screening, or has ever participated in a study with Imprime PGG or Betafectin®
7. Has donated or lost more than a unit of blood within 30 days of the last day of screening (Day -1)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2006-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
-To determine the safety of Imprime PGG when dosed as part of a standard 4-day regimen of G-CSF assessed via occurrence of adverse events and change from baseline in clinical laboratories, physical examination, vital signs and ECG | Prospective

SECONDARY OUTCOMES:
-To evaluate the progenitor cell mobilizing efficacy of Imprime PGG when dosed as part of a standard 4-day progenitor cell mobilizing regimen of G-CSF assessed through peripheral blood CD34+ cell counts | Prospective